CLINICAL TRIAL: NCT00559442
Title: Susceptibility to High Altitude Pulmonary Edema in Subjects With Increased Pulmonary Artery Pressure During Exercise in Normoxia and at Rest in Hypoxia
Brief Title: Susceptibility to High Altitude Pulmonary Edema in Subjects With Increased Hypoxic Pulmonary Vasoconstriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Internal Medicine VII, Sports Medicine, Medical Clinic, University Hospital of Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S-169/2007
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2007-11

CONDITIONS: High Altitude Pulmonary Edema
Keywords: high altitude pulmonary edema; hypoxic pulmonary vasoconstriction; right ventricular function; hypoxia
MeSH Terms: conditions — Altitude Sickness; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): high altitude exposure without prior acclimatization
  Interventions: Other: Altitude Exposure:

INTERVENTIONS:
Other: Altitude Exposure: — rapid ascent to Margherita Hut (4559 m) within 24 h

SUMMARY:
It has been shown, that subjects susceptible to high altitude pulmonary edema (HAPE)are characterized by an abnormal increase of pulmonary artery pressure at rest in hypoxia and during exercise in normoxia. This abnormal rise of pulmonary artery pressure has also been observed in about 10 % of otherwise healthy subjects without prior altitude exposure. The aim of the study is to investigate the susceptibility to HAPE in unacclimatized subjects with abnormal increase of pulmonary artery pressure at rest in hypoxia and during exercise in normoxia after rapid ascent to high altitude (4559 m).

ELIGIBILITY:
Inclusion Criteria:

* abnormal increase of pulmonary artery pressure at rest in hypoxia and during exercise in normoxia
* ability to climb Margherita Hut

Exclusion Criteria:

* Birth at or above 1500 m altitude
* any cardiovascular or pulmonary disease
* Infection disease
* Intake of drugs, in particular Acetazolamide, Nifedipine, corticosteroids or PDE-5-inhibitors.
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Frequency of HAPE after rapid ascent to 4559 m | during the 48 h stay at altitude

SECONDARY OUTCOMES:
Time course of pulmonary artery pressure | during the 48 h stay at altitude
Assessment of right ventricular function by echocardiography | during the 48 h stay at altitude

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Dehnert, MD, Principal Investigator — University Hospital Heidelberg; Ekkehard Grünig, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- Sports Medicine, University Hospital, Heidelberg, Germany

REFERENCES:
- [Derived] Dehnert C, Mereles D, Greiner S, Albers D, Scheurlen F, Zugel S, Bohm T, Vock P, Maggiorini M, Grunig E, Bartsch P. Exaggerated hypoxic pulmonary vasoconstriction without susceptibility to high altitude pulmonary edema. High Alt Med Biol. 2015 Mar;16(1):11-7. doi: 10.1089/ham.2014.1117. PMID 25803140